CLINICAL TRIAL: NCT04253795
Title: Comparative Study of Nonintubated Anesthesia With Laryngeal Mask Versus Intubated Anesthesia With Double Lumen Tube in Video-assisted Thoracic Surgery
Brief Title: Nonintubated Versus Intubated Anesthesia in Video-assisted Thoracic Surgery
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: not recruiting, awaiting for changes in IRB
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AntalyaTRH030
Record Dates: First submitted 2020-01-23; First posted 2020-02-05 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Intubation
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laryngeal mask group (Group 1) (Active Comparator): Laryngeal mask will be placed in the airway by the anesthesiologist. Lung isolation will be achieved with an artificial pneumothorax induced during opening the pleura, which resulted to the collapse of the nondependent lung with the patient's spontaneous breathing
  Interventions: Other: Laryngeal mask
- Double lumen tube Group (Group 2) (Active Comparator): After the correct position of double lumen tube will be determined, one lung ventilation will be started. Lung isolation will be achieved by deflation of the nondependent lung.
  Interventions: Other: double lumen tube

INTERVENTIONS:
Other: Laryngeal mask — After the laryngeal mask will be inserted lung isolation will be achieved with an artificial pneumothorax induced during opening the pleura, which resulted to the collapse of the nondependent lung with the patient's spontaneous breathing.
  Arms: Laryngeal mask group (Group 1)
Other: double lumen tube — After the one lung ventilation will be started, lung isolation will be achieved by deflation of the nondependent lung.
  Arms: Double lumen tube Group (Group 2)

SUMMARY:
The purpose of this study is to compare to the patients undergoing nonintubated general anesthesia with laryngeal mask and undergoing intubated general anesthesia with double-lumen endotracheal intubation in Video-assisted thoracic surgery (VATS).

DETAILED DESCRIPTION:
Although general anesthesia with double-lumen intubation is generally mandatory for Video-assisted thoracic surgery procedures intubation with double lumen tube is related to several risks. Nonintubated general anesthesia with laryngeal mask in patients with spontaneous breathing may be an alternative choice for minor VATS procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective minor VATS procedures will be enrolled the study

Exclusion Criteria:

* patients <18 years old,
* body mass index (BMI)>30 kg/m2,
* American Society Association (ASA) Class>3,
* heart failure (New York Heart Association class > II),
* a history of arrhythmia or treatment with antiarrhythmic drugs,
* bradycardia (heart rate (HR) <45 beats min1)
* atrioventricular block,
* hepatic or renal dysfunction,
* coagulopathy,
* asthma
* sleep apnea syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
difference in PaO2/FiO2 ratio at the end of the surgery | 1 hour
  PaO2/FiO2 ratio will be calculated for both groups at the end of the surgery

SECONDARY OUTCOMES:
Anesthesia time | 20 minutes
  Anesthesia time will be defined in minute as the time from starting electronically monitored in the operating room until the time the double lumen tube or laryngeal mask was correctly placed
Operating room time | 1 hour
  Operating room time will be defined in minute as the time from arrival to operating room until the patient will be transferred to the post anesthetic care unit.
Post anesthetic care unit (PACU) time | 30 minutes
  PACU time will be defined in minute as the time from arrival to the PACU until the patient was discharged to the ward.
Surgeon satisfaction | 10 minutes
  Surgeon will be asked to rate his satisfaction with the surgical conditions using a 4-point Likert scale (ie, "4: excellent", "3: good", "2: satisfactory", "1: unsatisfactory").
Patient satisfaction | 10 minutes
  Patient will be asked to rate his satisfaction using a 4-point Likert scale (ie, "4: excellent", "3: good", "2: satisfactory", "1: unsatisfactory").

CONTACTS AND LOCATIONS:
Overall Officials: Ali Sait Kavakli, M.D., Principal Investigator — Antalya Training and Research Hospital; Tayfun Sugur, M.D., Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Reseach Hospital Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)